CLINICAL TRIAL: NCT00134784
Title: [123I]ß-CIT and SPECT in Vivo Three Year Imaging Assessment of Dopamine Transporter Density in Subjects With Early Parkinson's Disease Participating in Earlier vs. Later Levodopa in Parkinson's Disease
Brief Title: Long-Term Dopamine Transporter Imaging and Clinical Assessment of Parkinson's Disease Progression
Acronym: ELLDOPA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institute for Neurodegenerative Disorders (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Kenneth Marek, MD, Principal Investigator, Institute for Neurodegenerative Disorders
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Elldopa
Record Dates: First submitted 2005-08-23; First posted 2005-08-25 (Estimated); Results first posted 2014-08-08 (Estimated); Last update posted 2014-08-08 (Estimated); Status verified 2014-07

CONDITIONS: Parkinson Disease
Keywords: parkinson; brain imaging
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Assess [123I]B-CIT SPECT imaging (Experimental): To assess[123I]B-CIT SPECT imaging in early Parkinson's disease subjects on placebo compared to early verses later Levodopa. Subjects on Levodopa 150mg/day, Levodopa 300 mg/day, and Levodopa 600 mg/day will be assessed.
  Interventions: Drug: [123I]B-CIT SPECT imaging

INTERVENTIONS:
Drug: [123I]B-CIT SPECT imaging — To assess [123I]B-CIT SPECT imaging
  Other Names: [123I]B-CIT

SUMMARY:
The purpose of this project is to assess the change in dopamine transporter density in Parkinson's disease subjects during a sixty month period including a nine month treatment trial of levodopa. Dopamine transporter will be assessed using [123I]ß-CIT SPECT (single photon emission computed tomography) imaging, a marker of dopamine terminal integrity and of clinical disease state.

DETAILED DESCRIPTION:
All subjects will be imaged at the Institute for Neurodegenerative Disorders.

Subjects will be evaluated sequentially with [123I]ß-CIT SPECT and standardized clinical rating scales during a sixty month period. The subjects involved in this study will have had [123I]ß-CIT and SPECT scans at baseline and return for scanning at week 40 following the start of their participation in the ELLDOPA study.

Before each SPECT procedure subjects will be tested to ensure eligibility for the study. They will also have a neurological evaluation including tests of motor function, thinking, memory and handwriting. Some of these tests will be given with the aid of a computer.

On the first day participants are injected with [123I]ß-CIT, an investigational radioactive material that localizes in the brain. Study participants will also have a thorough neurologic examination and standard neuropsychological testing, including testing of memory, concentration, abstraction and visual spatial functions.

Twenty-four hours later study participants return to the Institute for Neurodegenerative Disorders where an investigational scanning procedure will be used to obtain SPECT (single photon emission computed tomography) images of the brain.

ELIGIBILITY:
Inclusion Criteria:

* Prior participation in the study titled Dopamine Transporter Imaging Assessment of Parkinson's Disease Progression (DAMD17-99-1-9472) [123I] B-CIT and Spect in Vivo Imaging Assessment of Dopamine Transporter Density in Subjects With Early Parkinson's Disease Participating in Earlier Vs. Later Levodopa in Parkinson's Disease (ELLDOPA)].

Exclusion Criteria:

* Inability to sign informed consent and participate in all study procedures.
* Mini mental status exam < 25.
* Pregnancy

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2000-04; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth L Marek, MD, Principal Investigator — Institute for Neurodegenerative Disorders

REFERENCES:
- [Result] Fahn S, Oakes D, Shoulson I, Kieburtz K, Rudolph A, Lang A, Olanow CW, Tanner C, Marek K; Parkinson Study Group. Levodopa and the progression of Parkinson's disease. N Engl J Med. 2004 Dec 9;351(24):2498-508. doi: 10.1056/NEJMoa033447. PMID 15590952
- See also: Institute for Neurodegenerative Disorders — http://www.indd.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo group
- Levodopa 150mg/Day: Levodopa 150mg/day, [123I]ß-CIT and SPECT imaging
- Levodopa 300 mg/Day: Levodopa 300mg/day, [123I]ß-CIT and SPECT imaging
- Levodopa 600 mg/Day: Levodopa 600/day, [123I]ß-CIT and SPECT imaging
Period: Overall Study
Arm/Group | Placebo | Levodopa 150mg/Day | Levodopa 300 mg/Day | Levodopa 600 mg/Day
Started | 29 | 38 | 37 | 38
Completed | 27 | 36 | 35 | 37
Not Completed | 2 | 2 | 2 | 1
Not completed — Withdrawal by Subject | 2 | 2 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Placebo Group: Subjects on placebo
- Levodopa 150mg/Day: Subjects on 150mg/day of Levodopa
- Levodopa 300 mg/Day: Subjects on 300 mg/day of Levodopa
- Levodopa 600 mg/Day: Subjects on Levodopa 600 mg/day
- Total: Total of all reporting groups
Arm/Group | Placebo Group | Levodopa 150mg/Day | Levodopa 300 mg/Day | Levodopa 600 mg/Day | Total
Number analyzed (Participants) | 29 | 38 | 37 | 38 | 142
Age, Continuous [Mean (Standard Deviation); unit: years]
  Age of Subject in Years | 63.9 (10.5) | 64.5 (11.8) | 63.1 (10.2) | 62.3 (9.8) | 63.4 (10.6)
Sex/Gender, Customized [Number; unit: participants]
  Female | 7 | 15 | 8 | 11 | 41
  Male | 22 | 23 | 29 | 27 | 101

OUTCOME MEASURES:

1. Primary Outcome: Change in the Ratio of the Specific Striatal [123I]B-CIT Uptake to the Nondisplaceable Striatal [123I]B-CIT Uptake Between the Two Images
Description: The use of SPECT to measure striatal dopamine-transporter density with the use of [123I]B-CIT. Subjects underwent SPECT imaging just before the baseline visit and then again before the visit at week 40.
Time Frame: 40 weeks
Population: Per protocol
Measure: Mean (Standard Deviation); unit: percent change of B-CIT Uptake
Units Other Than Participants: B-CIT Uptake
Groups:
- Placebo Group: Participants receiving placebo
- Levodopa: Subjects on 150 mg/day of Levodopa
- Levodopa 2: Subjects on 300 mg/day of Levodopa
- Levodopa 3: Subjects on 600 mg/day of Levodopa
Arm/Group | Placebo Group | Levodopa | Levodopa 2 | Levodopa 3
Number analyzed (Participants) | 29 | 33 | 37 | 36
Number analyzed (B-CIT Uptake) | 29 | 33 | 37 | 36
percent change of B-CIT Uptake | -2.6 (11.3) | -4.7 (10.8) | -3.7 (9.1) | -6.9 (8.1)

ADVERSE EVENTS:
Groups:
- I123BCIT: [123I]ß CIT and SPECT imaging' .
Arm/Group | I123BCIT
Serious Adverse Events (participants affected / at risk) | 0/142
Other Adverse Events (participants affected / at risk) | 0/142

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes